CLINICAL TRIAL: NCT06035094
Title: An Exercise Intervention to Improve Overall Brain Health: PEDAL (Physical Education for an Active Lifestyle) Study
Brief Title: An Exercise Intervention to Improve Overall Brain Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pamela G Bowen PhD, CRNP, FNP-BC, BBA, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-300011511; 2027708 (Other Grant/Funding Number: McCance/ UAB)
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Brain Care Score; Exercise; Hypertension; BMI
Keywords: Brain health; brain care score; exercise; hypertension; overweight; obesity; BMI
MeSH Terms: conditions — Motor Activity; Hypertension; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Interval Training (HIIT) exercise group, (Experimental): Participants will be asked to exercise independently 4 days/week for 10 weeks, following a high intensity interval training (HIIT) protocol.
  Interventions: Behavioral: Exercise Intervention to improve overall Brain Health
- Moderate Intensity Training (MIT) exercise group (Experimental): Participants will be asked to exercise independently 4 days/week for 10 weeks, following a moderate intensity training (MIT) protocol.
  Interventions: Behavioral: Exercise Intervention to improve overall Brain Health
- Control exercise group (Active Comparator): Participants will be advised to follow the American Heart Association (AHA) guidelines on exercise.
  Interventions: Behavioral: Exercise Intervention to improve overall Brain Health

INTERVENTIONS:
Behavioral: Exercise Intervention to improve overall Brain Health — During each exercise session, the participant will be assigned to the HIIT or MIT exercise group and asked to ride the stationary bicycle for approximately 30-40 minutes, while wearing the heart rate monitor and recording the session on their smart phone application. For each exercise session, the Polar Beat application will record the time in each of four intensity "zones". The participant will receive training on how to use the outlined schedule during the initial supervised training session.

SUMMARY:
The goal of this clinical trial is to test the effects of 10 weeks of exercise on overall brain health, reduction in blood pressure, and the number of blood vessels in the back of the eyes in patients with hypertension and have a body mass index ≥ 25 kg/m2. The main question[s] it aims to answer are:

* To test the effect of moderate vs intensive exercise on Brain Care Score outcomes.
* To ascertain the differential impact of moderate vs high intensity exercise in reducing hypertension and its downstream effects.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with hypertension
* have a body mass index ≥ 25 kg/m2
* are between the ages of 35-65 years old
* access to a smart phone that allows installation of 2 two applications that record your workouts
* pass a fitness evaluation.

Exclusion Criteria:

* do not have hypertension
* weight over 300 lbs
* unable to pass the fitness evaluation
* BMI less than 25kg/m2

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-01-12 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
Improved overall Brain Care Score metric. | 10 weeks
  The score is based on lifestyle categories on a scale of 0-21 where 21 is best.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela G. Bowen, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No